CLINICAL TRIAL: NCT02092610
Title: Long Term Stability, Survival and Tolerability of a (Novel) Baha® Implant System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear Bone Anchored Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBAS5562
Record Dates: First submitted 2014-03-14; First posted 2014-03-20 (Estimated); Results first posted 2016-01-11 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Conductive Hearing Loss
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Implant BI300 (Active Comparator): The product was the standard titanium implant and abutment in the Baha system developed by Cochlear Bone Anchored Solutions AB. The implant is 3.75 mm wide and 4.0 mm long
  Interventions: Device: Standard Implant BI300
- Novel Implant BI300 (Experimental): The product was the novel titanium implant and abutment for the Baha system developed by Cochlear Bone Anchored Solutions AB. The novel implant is 4.5 mm wide and 4.0 mm long.
  Interventions: Device: Novel Implant BI300

INTERVENTIONS:
Device: Novel Implant BI300 — The Novel Implant BI300 was the new titanium implant and abutment for the Baha system developed by Cochlear Bone Anchored Solutions AB. The novel implant is 4.5 mm wide and 4.0 mm long.
  Arms: Novel Implant BI300
Device: Standard Implant BI300 — The Standard Implant BI300 was the standard titanium implant and abutment in the Baha system developed by Cochlear Bone Anchored Solutions AB. The implant is 3.75 mm wide and 4.0 mm long
  Arms: Standard Implant BI300

SUMMARY:
An international multicentre, open, comparative, parallel group, prospective clinical investigation with a single 5 year follow up visit.

DETAILED DESCRIPTION:
Two implant products, the standard implant and abutment and the novel implant and abutment, both developed by Cochlear Bone Anchored Solutions AB were tested in the CAG5173 clinical investigation that was completed in December 2012. The primary objective was to show superiority of the novel implant compared to standard implant in terms of implant stability quotient (ISQ) as as measured by resonance frequency analysis1. Results after 6 and 36 months after implantation showed that the new design, the novel implant and abutment, provided statistically significantly higher stability at the time of insertion and over time compared to the standard Baha implant2,3,4. In the investigation, sound processor fitting was performed from 6 weeks post-implantation. No reduction in implant stability following sound processor fitting was recorded, suggesting that it is safe to load the implant 6 weeks after implantation. The investigation also showed improved soft tissue outcomes, in terms of lower Holgers index5 scores for the novel implant and abutment compared to the standard implant and abutment.

After initiation of the 3-year CAG5173 investigation, Cochlear Bone Anchored Solutions AB launched the Cochlear Baha BIA300 Implant and Abutment, which in all critical aspects are identical to the novel implant used in the investigation.

The 36-month visit was the last visit of the investigation. Hence, no further visits were planned or scheduled for the subjects participating in that investigation.participating subjects. It is of clinical and scientific interest to evaluate the clinical performance and safety data of the implants in these subjects after an additional two-year period, in order to gain additional understanding of how implant stability and soft tissue status evolves over time with the two implant and abutment designs, and in order to evaluate long-term implant survival. No randomised controlled investigation of Baha implants with a 5-year follow-up has been conducted to date.

The rationale behind this clinical investigation is to collect long term stability, survival and tolerability data of a novel Baha implant system 5 years after implantation in a population that previously have been followed in a completed controlled investigation during a 3 year period. The collected data will enable comparison with the data gathered in the previous completed CAG5173 clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the CAG5173 investigation
* Signed informed consent

Exclusion Criteria:

* Unable to follow investigational procedure
* Any factor, at the discretion of the investigator, that is considered to contraindicate participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johan Blechert, M.Sc, Study Director — Cochlear Bone Anchored Solutions AB
Locations (4):
- Radboud University Medical Center, Nijmegen, Netherlands
- Sahlgrenska University Hospital, Gothenburg, Sweden
- United Kingdom (2):
  - Manchester Royal Infirmary, Manchester
  - Salford Royal hospital, Salford, Manchester

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Implant BI300 | Novel Implant BI300
Started | 25 | 52
Completed | 17 | 40
Not Completed | 8 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Implant BI300 | Novel Implant BI300 | Total
Number analyzed (Participants) | 17 | 40 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 21 | 27
  >=65 years | 11 | 19 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (9.4) | 55.4 (12.8) | 63.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 21 | 28
  Male | 10 | 19 | 29
Region of Enrollment [Number; unit: participants]
  Sweden | 2 | 7 | 9
  Netherlands | 11 | 26 | 37
  United Kingdom | 4 | 7 | 11
Implant stability measured by resonance frequence analysis [Mean (Standard Deviation); unit: ISQ scores] — The ISQ value ranges from 1 to 100, the higher value, the higher the implant stabilty.
  ISQ scores | 65.4 (3.2) | 70.1 (2.4) | 68.5 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Implant Stability
Description: To show superiority of the novel implant compared to standard implants regarding stability of the implants measured as ISQ values at the abutment level. The ISQ value ranges from 1 to 100, the higher ISQ value, the higher the implant stabilty. Mean AUC 0-60 months ISQ represents a weighted average of the implant stability during the 60 months from start of the CAG5173 study to the measurement in this study CBAS5562. The ISQ 5 years value represents the single ISQ measurment at 5 years.
Time Frame: At the single 60 months visit
Population: The 5 year follow up population consisted of the patients in the ITT population (all randomized subjects who received surgery) in the CAG5173 study who attended this study which was a 5-year follow up visit.
Measure: Mean (Standard Deviation); unit: ISQ scores
Arm/Group | Standard Implant BI300 | Novel Implant BI300
Number analyzed (Participants) | 17 | 40
ISQ scores
  AUC ISQ baseline to 5 years | 66.7 (3.4) | 71.6 (2.0)
  ISQ, 5 years | 67.4 (4.0) | 72.1 (2.2)

2. Secondary Outcome: Longterm Survival of Implant
Description: To compare the long term survival of the novel implant and abutment and the standard implant and abutment in the Baha system.
  All patients will be asked if they have experienced any implant osseointegration problems which would have made the implant to get loose. The time from implant implantation until implant loss or removal will be collected. In case of implant removal, reason for removal shall be recorded.
Time Frame: At the single 60 months visit
Population: Survival population, all patients in the ITT population in the original study CAG5173 (all randomized patients who get surgery).
Measure: Number; unit: % survival rate of implants
Arm/Group | Standard Implant BI300 | Novel Implant BI300
Number analyzed (Participants) | 25 | 52
% survival rate of implants
  Survival rate including explants | 90.0 | 93.92
  Survival rate excluding explants | 95.0 | 95.8

3. Secondary Outcome: Soft Tissue Status
Description: To evaluate the status of the soft tissue at the implant site.
  The scale Holgers Index 4 is designed to capture signs and symptoms of inflammation or infection at the site of implantation. The scale should be completed at the visit.
  The scale consists of the following steps:
  0. No irritation. Epidermal debris removed, if present
  1. Slight redness. Local temporary treatment, if needed
  2. Red and slightly moist tissue. No granulation formation, local treatment and extra controls as indicated
  3. Reddish and moist; sometimes granulations tissue, revision surgery is indicated
  4. Removal of the abutment/implant necessary due to infection R. Removal of abutment/implant for reasons not related to skin problems
Time Frame: At the single 60 months visit
Population: Five year follow up population
Measure: Number; unit: % of participants
Arm/Group | Standard Implant BI300 | Novel Implant BI300
Number analyzed (Participants) | 17 | 40
% of participants
  No irritation | 52.9 | 90.0
  Slight redness | 23.5 | 7.5
  Red and slightly moist tissue | 23.5 | 2.5
  Reddish and moist | 0 | 0
  Removal of abutment is necessary due to infection | 0 | 0

4. Secondary Outcome: Implant Survival
Time Frame: 60 months
Population: These data are already presented in the "Longterm Survival of Implant" section.
Arm/Group | Standard Implant BI300 | Novel Implant BI300
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Standard Implant BI300 | Novel Implant BI300
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/40
Other Adverse Events (participants affected / at risk) | 0/17 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days